CLINICAL TRIAL: NCT04755049
Title: The Chinese Version of the American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form Questionnaire, Patient Self-report Section: A Cross-cultural Adaptation and Validation Study
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Kai-Lan Hsu, Attending physician, National Cheng-Kung University Hospital
Other Study IDs: A-ER-109-163
Record Dates: First submitted 2021-02-06; First posted 2021-02-15 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: The Chinese version of the American Shoulder and Elbow Surgeons standardized shoulder assessment form questionnaire — The Chinese version of the American Shoulder and Elbow Surgeons standardized shoulder assessment form questionnaire

SUMMARY:
Background: The patient self-report section of the American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form (ASESp) is one of the most validated and reliable assessment tools. This study aimed to establish a validated Chinese version of ASESp (ASESp-CH).

Methods: A clinical prospective study was performed. Following the guidelines of forward-backward translation and cross-cultural adaptation, a Chinese version of ASESp was established. Patients older than 18 years with shoulder disorders were included. Patients who could not complete test-retest questionnaires within the interval of 7-30 days and patients who received interventions were excluded. Intraclass correlation (ICC) was calculated for test- retest reliability, whereas internal consistency was determined by Cronbach value. Construct validity was evaluated by comparing the corresponding domains between the ASESp-CH and a validated Chinese version of 36-Item Short Form Health Survey (SF-36).

ELIGIBILITY:
Inclusion Criteria:

* [1] patients' age ≥ 18 years
* [2] patients with clear insights
* [3] patients with any shoulder disorders
* [4] patients who are able to speak and write in Chinese
* [5] patients who completed the questionnaires twice at an interval of 7 days to 30 days.

Exclusion Criteria:

* [1] the patient could not complete all of ASESp-CH and SF-36 questionnaires
* [2] the test-retest interval was less than 7 days or more than 30 days
* [3] the patient received interventional procedures, such as shoulder injections or surgery, during the test-retest interval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with any shoulder disorders
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
The Chinese version of the American Shoulder and Elbow Surgeons standardized shoulder assessment form questionnaire | The questionaire was completed at 7 days before the index surgery.
  American Shoulder and Elbow Surgeons (ASES) Assessment Form, ranging from 0-100. The higher score indicates better shoulder function.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tie TA, Hong CK, Chua I, Kuan FC, Su WR, Hsu KL. The Chinese version of the American shoulder and elbow surgeons standardized shoulder assessment form questionnaire, patient self-report section: a cross-cultural adaptation and validation study. BMC Musculoskelet Disord. 2021 Apr 24;22(1):382. doi: 10.1186/s12891-021-04255-z. PMID 33894753